CLINICAL TRIAL: NCT04478188
Title: The Use of PV Loop Analysis to Optimize Cardiogenic Shock and Device Management
Brief Title: Pressure Volume Loop
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Danny Ramzy, Director, Robotic Cardiac Surgery, Principal Investigator, Assosiate Professor of Surgery, Cedars-Sinai Medical Center
Other Study IDs: 00000164
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Cardiogenic Shock; Decompensated Heart Failure
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiogenic Shock Patients Needing TMCS: Heart failure patients who undergo TMCS insertion for acute decompensated heart failure and cardiogenic shock.
  Interventions: Other: Measuring Pressure Volume Loop Pre and Post Device Placement

INTERVENTIONS:
Other: Measuring Pressure Volume Loop Pre and Post Device Placement — To measure simultaneous pressure and volume of the heart (pressure volumes loops) before and after ventricular assist device placement for cardiogenic shock (a severe form of heart failure) and before and after device removal.

SUMMARY:
The investigators are doing this study and medical record review to measure simultaneous pressure and volume of the heart called pressure volumes loops before and after ventricular assist device placement for cardiogenic shock ( a severe form of heart failure). Standard of care measurements will be the sole measure of clinical determination. The investigators are measuring these PV loops to help determine which patients heart have recovered and can have the ventricular assist device removed. The investigators are also using the PV loop to indicate/correlate with certain outcomes to predict the need for LVAD patients to require additional support in the form of a right ventricular assist device. The medical record review will be performed pre-operatively, intra-operatively, and post-operatively until the day of discharge.

DETAILED DESCRIPTION:
Cardiogenic shock (CS) represents a high risk population that is at risk for both in-hospital mortality and readmission following discharge. CS can be either left ventricular (LV) or right ventricular (RV) or of biventricular (BiV) origin. Even in patients with CS treated with an invasive approach (cardiac catheterization, angioplasty, and coronary bypass surgery), in-hospital mortality approaches 50%. Other causes of CS mainly include severe decline in underlying systolic function (from non-ischemic causes such as sepsis, stress, and progression of systolic left ventricular dysfunction among others), arrhythmias, and mechanical cardiac complications. Cardiogenic shock in the absence of acute myocardial infarction (AMI) (non-AMI CS) is excluded from most studies including randomized trials and remains largely understudied. For many years, the intra-aortic balloon pump was thought to be helpful in improving outcomes in cardiogenic shock. However, the landmark randomized, controlled IABP-SHOCK II trial, published in 2012, and concluded that the use of intra-aortic balloon counter pulsation did not significantly reduce mortality in patients with cardiogenic shock complicating acute myocardial infarction. This led investigators to search for alternate temporary mechanical circulatory support systems that might prove effective in reducing mortality in cardiogenic shock. One such system is the Impella 5.0 and Impella RP devices. The Impella 5.0 pump in a temporary continuous flow pump approved for hemodynamic support for left ventricular shock CS patient and the Impella RP for right ventricular shock. The other system is the Tandem heart pump. The investigators utilize the Impella and the tandem pump for AMI CS and non-ischemic CS. The device is implanted for bridge to recovery, bridge to transplant and as a bridge to durable device. The investigators have discovered that recovery rates following AMI shock are significantly improved with the Impellaand tandem heart pumps however; identifying which patient recovers remains a mystery. Adequate parameters do not exist.

Patients who we are unable to recover are transitioned to a durable continuous flow left ventricular assist devices (CF-LVAD) which are an effective alternative to heart transplant, but are not risk-free: among the other effects, right ventricle (RV) hemodynamics are significantly altered by the LVAD implantation. In fact, RV failure occurs in 5% of patients with implanted CF-LVADs, and leads to a 6-fold increase in the risk of death. Moreover, RV failure is a major contributing factor in prolonged hospitalizations, and is associated with a higher risk of bleeding, renal failure, and hypotension. Currently, predictors of RV failure in patients undergoing LVAD implantation are based entirely on retrospective case series, often evaluating cohorts of patients with outdated classes of pulsatile-flow LVADs.Furthermore, right ventricular failure (RVF) still results as the major cause of morbidity and mortality after LVAD implantation. Despite overall improved outcomes and lower rates of RVF with the use of the newer, LVAD over pulsatile-flow devices, and development of clinical prediction scores to facilitate preoperative identification of patients at risk for RVF after implantation remains elusive. RVF occurs in 13% to 40% of continuous-flow device. The ability to predict the development of RV failure post LVAD implantation would significantly improve outcomes as these patients would either have planned RVAD implantation or receive a total artificial heart implantation.

ELIGIBILITY:
Inclusion Criteria:

All cardiogenic shock patients requiring temporary mechanical circulatory support (TMCS) (Impella, Tandem heart and ECMO). Age >=18

-

Exclusion Criteria:

* Age <18, All patients requiring ECRP
* Patients with a Mechanical Aortic Valve
* Patients with Left Ventricular Thrombus

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All cardiogenic shock patients requiring mechanical circulatory support devices can be enrolled in the study. The patients chart will be examined for possible exclusion by the PI or implanting surgeon who is also a co-investigator.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Ventricular Pressure Volume Loop Analysis | Up to 90 days
  Three Load independent Parameters will be measured and analyzed at three different time points. Pre, post implant and at explant

SECONDARY OUTCOMES:
Survival and device explant rate | 1 year
  Measurement of the proportion of patients that were able to be weaned off the device and percent survival

CONTACTS AND LOCATIONS:
Overall Officials: Danny Ramzy, MD, Principal Investigator — Physician
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time there are no plans to share individual participant data with other researchers